CLINICAL TRIAL: NCT00488007
Title: Clinical Trial on Cognitive, Behavioural, Quality of Life and Medico-economic Benefits of Hearing Aids in Alzheimer Disease Patients Suffering From Presbycusis
Brief Title: Clinical Trial on Alzheimer Disease, Presbycusis and Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006.414
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease; Presbycusis
Keywords: Alzheimer disease; Cognitive impairment; Sensorineural hearing loss; Hearing aids
MeSH Terms: conditions — Alzheimer Disease; Presbycusis; Cognitive Dysfunction; Hearing Loss, Sensorineural

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Hearing aids (Experimental): Active
  Interventions: Device: Hearing aids used : PHONAK Savia and Valeo
- Inactive Hearing aids (Placebo Comparator): Hearing aids turned off
  Interventions: Device: Hearing aids used : PHONAK Savia and Valeo

INTERVENTIONS:
Device: Hearing aids used : PHONAK Savia and Valeo — 5 hours per day during the first 6 months (active or inactive upon randomization) 5 hours per day during the last 6 months (active)

SUMMARY:
This is a 12-months' randomized clinical trial that aims at studying the benefit of bilateral hearing aids in hearing impaired patients suffering from a slight to moderate stage Alzheimer disease.

The benefit of this intervention will be studied in the cognitive, behavioural, quality of life and economic fields.

2groups are involved in this trial: Intervention group: 12 months' treatment with active hearing aids, fitted hearing impairment Control group: 6 months' treatment with placebo hearing aids, followed with 6 months' active hearing aids, fitted hearing impairment

ELIGIBILITY:
Inclusion Criteria:

* > 65 year-old
* Medical diagnosis of Alzheimer disease
* 15 ≤ MMSE ≤ 25
* No hearing aids in the last 2 years
* Motivated caregiver living with the patient
* Sensorineural hearing loss

Exclusion Criteria:

* Beginning of an anticholinesterasic treatment in the last 6 months
* Change in the anticholinesterasic treatment in the last 2 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-05; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cognitive benefit evaluated thanks to the ADAS-Cog scale | Times of measurements: 0, 6th and 12th month

SECONDARY OUTCOMES:
Cognitive scales: MMSE, Grober and Buschke, Digit symbol test | 0, 6th and 12th month
Behavioural scales: IADL, NPI | 1st week, 3rd 6th 9th and 12th month
Quality of life scales: Zarit scale and ADRQL | Zarit scale(every 2 months during the study time), ADRQL (0, 6th and 12th month)
Consumption questionnaire | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Marc BONNEFOY, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Xavier PERROT, Lyon, France

REFERENCES:
- [Result] Adrait A, Perrot X, Nguyen MF, Gueugnon M, Petitot C, Collet L, Roux A, Bonnefoy M; ADPHA study group. Do Hearing Aids Influence Behavioral and Psychological Symptoms of Dementia and Quality of Life in Hearing Impaired Alzheimer's Disease Patients and Their Caregivers? J Alzheimers Dis. 2017;58(1):109-121. doi: 10.3233/JAD-160792. PMID 28269769
- [Result] Nguyen MF, Bonnefoy M, Adrait A, Gueugnon M, Petitot C, Collet L, Roux A, Perrot X; ADPHA study group. Efficacy of Hearing Aids on the Cognitive Status of Patients with Alzheimer's Disease and Hearing Loss: A Multicenter Controlled Randomized Trial. J Alzheimers Dis. 2017;58(1):123-137. doi: 10.3233/JAD-160793. PMID 28387664